CLINICAL TRIAL: NCT00887133
Title: Effectiveness of Western Medicine Outpatient Consultations in Primary Care - A Comparison With Chinese Medicine Consultations
Brief Title: Effectiveness of Western Medicine Outpatient Consultations in Primary Care
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Tung Wah Group of Hospitals (Other)
Responsible Party: Cindy L. K. Lam, Family Medicine Unit, The University of Hong Kong
Other Study IDs: HKCTR-477
Record Dates: First submitted 2009-04-06; First posted 2009-04-23 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Musculoskeletal Problem; Respiratory Problem; Gastrointestinal Problem; All Primary Care Problem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients consulting Western Medicine outpatient clinics for a new episode of illness

SUMMARY:
Background:

Primary care plays an important role in health care delivery, but there is little research on its effectiveness. Western medicine is the most widely used and Traditional Chinese medicine (TCM) is gaining popularity. The investigators recent study showed that TCM consultations at the TWH were effective in improving the quality of life of patients in primary care. The aim of the present study is to evaluate the effectiveness of Western Medicine (WM) in primary care for comparison with the effectiveness of TCM consultations, so that policy makers and the public can be better informed.

Objectives:

To evaluate whether WM consultation can significantly improve the quality of life of patients in primary care and to find out whether there is any difference in the effectiveness of WM and TCM, overall and for different health problems.

Design, Setting & Subjects:

A prospective study on 700 patients recruited from the TWH and the Ap Lei Chau primary care outpatient clinics (OPC) in Hong Kong.

Methods:

All patients consulting for a new episode of illness at the study OPC will be recruited if they meet the selection criteria and consent to participate. Each patient will be asked to complete a structured questionnaire on socio-demography, morbidity and service utilization, the Hong Kong version of the Chinese Quality of Life instrument (ChQOL-HK), the Chinese (Hong Kong) SF-36 (SF-36-HK) and the PEI-2 before the consultation. Each subject will be followed up two weeks later either at the clinic or by telephone to complete the ChQOL-HK and the SF-36-HK again together with the Patient Enablement Instrument (PEI), the Global Rating Scale (GRS) on change of the condition, and a questionnaire on service utilization

Outcome Measures and Data Analysis:

The primary outcome measures are the changes in ChQOL-HK and SF-36-HK scores after the consultation. The GRS and PEI scores will be secondary outcomes. The ChQOL -HK and SF-36-HK scores will be correlated with the the GRS and PEI. Multivariate regressions will be carried out to identify factors that are associated with effectiveness. The outcomes will be compared with those obtained from the previous study on the TCM primary care clinics.

Results:

This is the first study in Hong Kong to evaluate the effectiveness of WM in primary care with a validated generic outcome measure, HRQOL. It will provide information on the benefit and limitations of WM, and allow a direct comparison between WM and TCM.

DETAILED DESCRIPTION:
Primary health care serves every person and manages over 90% of the illnesses. The Hospital Authority public general and family medicine outpatient clinics provide about 11 million attendances each year, which is the major source of health care for the elderly and low-income population. The effectiveness of primary care has profound impact on the health of the population as well as the demand on expensive secondary care. Western medicine (WM) is the most commonly used type of primary care but 50 to 60% of people also consult Traditional Chinese medicine (TCM) in Hong Kong. The two types of medicine are often used sequentially or concurrently. There is a constant debate on whether WM or TCM is more effective, but few if any, comparative data are available. Few studies have investigated patient satisfaction with the public primary care clinics but none has investigated the effectiveness of care. A proper evaluation with a valid outcome measure will help to inform the public and policy makers on the benefit and limitations of the different primary care.

The evaluation of the effectiveness of a health service needs to use appropriate outcome measures. Health-related quality of life (HRQOL) with an emphasis on subjective perception of well-being and function is probably the most suitable outcome measure in primary care because most of the health problems are functional rather than pathological. The other advantage of HRQOL is that it is generic in that the same standard measure can be applied to different types of patients, illnesses and medical services.

Our previous study showed that all patients had significant improvements in their HRQOL after TCM consultations at the different (internal medicine, bone-setting and acupuncture) primary care outpatient clinics in Tung Wah Hospital. We would like to carry out a study to evaluate the effectiveness of WM in improving the HRQOL of patients attending the WM general outpatient clinic of the TWH and another public primary care clinic. To the best of our knowledge, this is the first study to evaluate the effectiveness of care of the public primary care service. The results will allow a direct comparison between WM and TCM, overall and for different illnesses, which can help to determine their respective roles in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient consulted the primary care clinic for the first time or a new episode of illness
* Gave consent to take part in the study

Exclusion Criteria:

* The visit to the primary care clinic was a follow up consultation
* Unable to communicate in Cantonese or Chinese
* Too ill to complete an interview
* Refused to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 1469 (Actual)
Dates: Start 2005-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The change in ChQOL-HK and SF-36-HK Scores, from baseline to 2 weeks The Chinese Quality of Life Questionnaire (ChQOL) The Hong Kong version of the Chinese Quality of Life Questionnaire (ChQOL - HK) was adapte | day 0 and day 14

SECONDARY OUTCOMES:
The Patient enablement instrument score and the Global rating of change score | day 0 and day 14

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L K Lam, MD, Principal Investigator — Family Medicine Unit, Faculty of Medicine, HKU
Locations (1):
- Two General Outpatient Clinics, Hong Kong, Hong Kong, China